CLINICAL TRIAL: NCT06471439
Title: An Investigation of Different Type Single Limb Exercise Training Effects on Functional Capacity, Arterial Stifness, Muscle Activation and Quality of Life in Chronic Obstructive Pulmonary Disease
Brief Title: An Investigation of Different Type Single Limb Exercise Training Effects in Copd
Acronym: COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Kocaaga, principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA-22104
Record Dates: First submitted 2024-05-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Exercise
Keywords: Chronic Obstructive Pulmonary Disease; Single Limb exercise; resistance training; continous exercise training; high intensity exercise training
MeSH Terms: conditions — Motor Activity; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: three different type one leg exercise intervention are apllied in patients with copd
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single leg resistance exercise intervantion in COPD (Active Comparator): single leg resistance exercise intervantion in COPD will be perfomed at six weeks
  Interventions: Other: single leg exercise intervantion in COPD
- single leg continous exercise intervantion in COPD (Active Comparator): single leg continous exercise intervantion in COPD will be perfomed at six weeks
  Interventions: Other: single leg exercise intervantion in COPD
- single leg high intensity exercise intervantion in COPD (Active Comparator): single leg high intensity exercise intervantion in COPD will be perfomed at six weeks
  Interventions: Other: single leg exercise intervantion in COPD

INTERVENTIONS:
Other: single leg exercise intervantion in COPD — single leg exercise intervantions
  1. high intensity interval training
  2. continous exercise training
  3. resistance exercise training
  Other Names: single leg exercise intervantion

SUMMARY:
COPD presents not only respiratory symtoms but also vascular or muscle dysfunction. Exercise limitation is observed in COPD. Especially, decreased exercise performance related to vascular and fatique in quadriceps muscle. Exercise training is important for aerobic performance increasing. Generally results show exercise training with both lower limb. Increaed arterial stiffness and fatigue are observed in COPD. One leg exercise training result is not enough to highlight these parameters.

Three types single leg exercise intervantion will be applied. Exercise capacity, muscle strength, lung function, electromyography, lactate and quality of life will be measured.

DETAILED DESCRIPTION:
Three types single leg exercise intervantion will applied to COPD patients that devided three groups. One leg continuous exercise training will be aplied to one group. One leg HIIT exercise training will be aplied to other group. One leg resistance exercise training will be aplied to the last group.

Exercise capacity and muscle strength are assesed. Lung function is measured. Electormyography is recorded. Lactate and quality of life are measured.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients that applied to physiotherapy
* Cooperation for tests
* without severe ortopedical and neurological disease
* without severe cardiovascular disease
* To volunteer for the study.

Exclusion Criteria:

* have an acute exacerbation or having exacerbation at last month
* hypoxemia (PaO2<55mmHg)
* no cooperated to test without volunteer to study having ortophedical and neurological diesase that affecting of tests severe cardiovascular disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
six minute walk test | pre-intervention
  six minute walk test in meter

SECONDARY OUTCOMES:
cardiopulmonary exercise test | beginning day 2
  VO2 as ml/kg/min will be recorded from incremental cycle cpet test
one leg cardiopulmonary exercise test | beginning, day 3
  VO2 as ml/kg/min will be recorded from incremental cycle cpet test
quadriceps muscle strength assesing (repeated measeure) | beginning day 1 and last day
  quadriceps muscle 10 repeated max muscle strength will be recorded at kilogram,
isometrics quadriceps muscle strength assesing | beginning day 1 and last day
  quadriceps muscle isometric muscle strength will be recorded at kilogram
lung function | beginning day 1 and last day
  FEV1/FVC ratio in %
quality of life assesing | beginning day 1 and last day
  total score in 0-100 range
arterial stiffness | beginning day 2 and last day
  total vascular resitance, augmentation index @ 75 and pulse wave velocity wil be determined arterial stiffness
lactate measurement | beginning day 2 and last day
  lactate in mmol
electromyography measurement | beginning day 2 and last day
  precentage of maximum volunteer contraction) %MVC values will be presented muscle fatigue (median frequence) and activation will be shown electromyograpy (EMG)

CONTACTS AND LOCATIONS:
Overall Officials: elif kocaaga, ms, Principal Investigator — Hacettepe University
Locations (1):
- Elif Kocaaga, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Dolmage TE, Goldstein RS. Effects of one-legged exercise training of patients with COPD. Chest. 2008 Feb;133(2):370-6. doi: 10.1378/chest.07-1423. Epub 2007 Oct 9. PMID 17925417
- [Background] Evans RA, Dolmage TE, Mangovski-Alzamora S, Romano J, O'Brien L, Brooks D, Goldstein RS. One-Legged Cycle Training for Chronic Obstructive Pulmonary Disease. A Pragmatic Study of Implementation to Pulmonary Rehabilitation. Ann Am Thorac Soc. 2015 Oct;12(10):1490-7. doi: 10.1513/AnnalsATS.201504-231OC. PMID 26291542
- [Background] MacInnis MJ, Morris N, Sonne MW, Zuniga AF, Keir PJ, Potvin JR, Gibala MJ. Physiological responses to incremental, interval, and continuous counterweighted single-leg and double-leg cycling at the same relative intensities. Eur J Appl Physiol. 2017 Jul;117(7):1423-1435. doi: 10.1007/s00421-017-3635-8. Epub 2017 May 11. PMID 28497384